CLINICAL TRIAL: NCT00856427
Title: Implantation of Markers for the Radiotherapy of Lung Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11284; HM11284 (Other: VCU IRB); CDR0000630623 (Registry Identifier: PDQ (Physician Data Query)); NCI-2013-00512 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IA non-small cell lung cancer; stage IB non-small cell lung cancer; stage IIA non-small cell lung cancer; stage IIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (Experimental): Patients undergo implantation of radio-opaque markers into the primary lesion and affected lymph nodes by bronchoscopy. Patients then undergo routine 4D CT, 4D CBCT, fluoroscopy, and x-ray imaging during standard stereotactic radiation therapy (early stage tumors) or conventionally fractionated radiation therapy (advanced stage tumors).
  Interventions: Radiation: radiation therapy treatment planning/simulation; Procedure: implanted fiducial-based imaging

INTERVENTIONS:
Radiation: radiation therapy treatment planning/simulation — Undergo implantation of radio-opaque markers
Procedure: implanted fiducial-based imaging — Undergo implantation of radio-opaque markers

SUMMARY:
This clinical trial studies imaging markers in planning radiation therapy in patients with lung cancer. Implanting markers in the tumor that can be seen using imaging procedures during radiation therapy may allow x-rays to be sent directly to the tumor and cause less damage to normal tissue.

DETAILED DESCRIPTION:
OBJECTIVES:

* To acquire experience in the marker implantation process for mediastinal lymph nodes and primary lung tumors in patients with stage I-IIIB non-small cell lung cancer.
* To characterize the potential side effects involved in the use of markers in these patients.
* To analyze the positional stability of lung markers in these patients over a radiotherapy series.
* To acquire experience in the use of markers for treatment planning and radiotherapy in these patients.

OUTLINE: Patients undergo implantation of ≥ 1 small radio-opaque Visicoil™ marker into or close to the primary lesion and affected lymph nodes by bronchoscopy. Patients then undergo x-rays to document marker location, detect potentially dropped markers, and diagnose operation-related side effects (i.e., pneumothorax). After marker implantation, patients undergo stereotactic or conventionally fractionated radiotherapy for 30-33 daily fractions.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer

  * Stage I-IIIB disease
* No prior surgical tumor resection
* Respiration-induced tumor motion > 5 mm
* Recruited by attending physician or research nurse at the Medical College of Virginia Hospitals

PATIENT CHARACTERISTICS:

* Not pregnant
* No insufficient lung function or other parameters prohibiting a bronchoscopy
* Not a prisoner or institutionalized

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent chemotherapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of dropped markers | up to 5 years
Marker misplacements | up to 5 years
Implantation-related side effects | up to 5 years
Visibility of markers on CT and x-rays | up to 5 years
Positional reliability of markers | Up to 5 years
Usability for patient treatment | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Weiss, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia, United States